CLINICAL TRIAL: NCT00008099
Title: Phase I Dose Escalation Trial of a 100 aa Synthetic Mucin Peptide Admixed With SB-AS2 as Adjuvant in Locally Advanced and Resected Pancreatic Cancer
Brief Title: Vaccine Therapy in Treating Patients With Resected or Locally Advanced Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Herbert J. Zeh, III MD, FACS, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCI-97-046; CDR0000068375 (Registry Identifier: PDQ (Physician Data Query)); PCI-IRB-970871; NCI-G00-1888
Record Dates: First submitted 2001-01-06; First posted 2004-05-04 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: MUC1 antigen/SB AS-2

SUMMARY:
RATIONALE: Vaccines may help the body build an effective immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with resected or locally advanced unresectable pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and toxicity of vaccination with MUC-1 antigen and immunologic adjuvant SB AS-2 in patients with resected or locally advanced unresectable pancreatic cancer. II. Determine the maximum tolerated dose and/or recommended phase II dose of MUC-1 antigen in this patient population. III. Determine the qualitative and quantitative tumor response to this treatment in these patients. IV. Determine the disease-free survival in resected patients, progression-free survival in locally advanced unresectable patients, and overall survival in all patients receiving this treatment.

OUTLINE: This is a dose escalation study of MUC-1 antigen. Patients receive vaccination with MUC-1 antigen and immunologic adjuvant SB AS-2 intramuscularly on day 1. Treatment repeats every 3 weeks for a total of 3 courses in the absence of disease progression or unacceptable toxicity. Beginning 1 year after the last vaccination, patients without recurrent disease may receive booster vaccines annually. Cohorts of 4 to 8 patients receive escalating doses of MUC-1 antigen until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 4 or 2 of 8 patients experience dose-limiting toxicity. Patients are followed at 2 weeks.

PROJECTED ACCRUAL: A total of 15-20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed resected or locally advanced unresectable pancreatic cancer No metastases

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-2 Life expectancy: At least 4 months Hematopoietic: WBC greater than 3,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective double barrier contraception 1 week before, during, and for at least 2 weeks after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: No concurrent glucocorticosteroids Radiotherapy: No prior radiotherapy Surgery: At least 3 weeks since prior resection of pancreatic cancer Other: No concurrent non-steroidal anti-inflammatory drugs (NSAIDs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1998-05; Primary Completion 2001-03 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Disease Recurrence | 1-2 years

SECONDARY OUTCOMES:
Overall Survival | 2-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh K. Ramanathan, MD, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States